CLINICAL TRIAL: NCT04916639
Title: Seawater Nasal Wash to Relieve COVID-19 Nasal Symptoms and Reduce SARS-CoV-2 Viral Load.
Acronym: SeaCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire de la Mer (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SeaCare
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: SARS-CoV2 Infection (COVID-19); URTI - Viral Upper Respiratory Tract Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Physiomer®, undiluted seawater nasal spray
  Interventions: Device: Device: Physiomer undiluted seawater nasal spray
- control group (No Intervention)

INTERVENTIONS:
Device: Device: Physiomer undiluted seawater nasal spray — In this study, subjects are asked to adhere to the following dosage during the 3 weeks of the study:
  * Nasal wash four times every day
  * These washes are to be carried out in each nostril
  * By continuously pressing the spray for 3 seconds in each nostril
  * Subjects are recommended to distribute the 4 nasal washes as follows:
    * 1st : morning
    * 2nd : midday
    * 3rd : afternoon
    * 4th : evening Subjects will be instructed to maintain daily nasal wash over the 3 weeks study period even in case of earlier nasal symptoms resolution, in order to assess the impact of nasal wash on viral load and other symptoms.
  Arms: Active group

SUMMARY:
Prospective, randomized, controlled, multicenter, parallel clinical trial to assess the efficacy of seawater nasal wash to relieve COVID-19 and URTIs nasal symptoms and reduce intranasal viral load in subjects with mild to moderate COVID-19 disease and URTIs.

DETAILED DESCRIPTION:
SARS-CoV-2 coronavirus enters into the human body mainly through the angiotensin converting enzyme 2 (ACE2) and transmembrane protease serine 2 (TMPRSS2) nasal epithelial cells. Like many other airborne viral diseases, penetration into the upper respiratory tract (URT) is the first step of the infection. Once SARS-CoV-2 enters the host via the respiratory tract, airway and alveolar epithelial cells, vascular endothelial cells and alveolar macrophages are among the first targets of viral entry. Several studies have reported that the viral loads in the upper respiratory tract (URT) peak at the time of, or early after, onset of symptoms. Higher virus load in upper respiratory tract (URT) also induces a higher overall SARS-CoV-2 household secondary attack rate.

Nasal saline irrigations are frequently prescribed for both prevention and treatment of upper respiratory tract infections (URTIs). Nasal wash provides mechanical cleansing of mucus, crust, cell debris and various air contaminants including pathogens (virus and bacteria). It enhances mucociliary clearance and reduces the mucus contact time of airborne elements. The effectiveness of nasal lavage has been shown to reduce the duration of infectious episodes and relieve symptoms of upper respiratory tract infections (URTIs) caused by various respiratory viruses including coronaviruses. Preliminary data showed that daily nasal wash can significantly reduce symptom duration in subjects with mild and moderate forms of COVID-19.

The sponsor hypothesized that the daily use of seawater nasal wash in subjects with mild to moderate forms of COVID-19 or URTIs:

* Would relieve nasal symptoms caused by SARS-CoV-2 and URTIs virus, including nasal obstruction and rhinorrhea.
* Would reduce the intranasal viral load by mechanical evacuation of nasal secretions containing the viruses, and by reducing the contact time between the viruses and the nasal mucosa.

The main objective of this study is to evaluate the effectiveness of Physiomer®, an undiluted isotonic seawater nasal spray, on reducing the duration of nasal symptoms (nasal obstruction or rhinorrhea) in subjects with mild to moderate COVID-19 and URTIs.

The study will take place in France among adults subjects who developed nasal obstruction and rhinorrhea no more than 48 hours before study inclusion. Subjects will be randomized into one of two study groups: control group or nasal wash group. Subjects in the nasal wash group will be asked to perform daily nasal wash for a 3 weeks period with Physiomer®, a 100% seawater isotonic nasal spray. Subjects in both groups will complete daily online questionnaires for a 3 weeks period. In order to follow the evolution of intra-nasal viral load, 4 naso-pharyngeal swabs will be collected at home by a nurse.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years) with self-reported nasal obstruction and/or rhinorrhea ≤48 hours due to COVID-19 or URTIs
* Willing to have regular nasopharyngeal swabs as per protocol
* Subjects agreeing to follow the study requirements during the whole study period
* Subject affiliated to social security
* Subject able to understand verbal and written local language and in capacity to fill-in questionnaire by himself

Exclusion Criteria:

* Age over 65 years
* Subjects requiring hospitalization
* Subjects with severe COVID-19 symptoms
* Inability or unwillingness to perform saline irrigations
* subjects who have performed nasal wash in the previous week including the day of inclusion
* Requirement to take regular medications administered by nasal route (topical treatment such as corticosteroids, antihistaminics, vasoconstrictors, inhalation)
* Subjects intending to undergo nasal surgery during the study period or who underwent nasal surgery in the 3 previous months.
* Pregnancy or breastfeeding
* Cardiovascular pathologies: history of stroke, history of coronary artery disease, history of cardiac surgery, NYHA stage III or IV heart failure;
* Asthma (requiring treatment)
* Chronic pulmonary / respiratory pathology (cystic fibrosis, obstructive pulmonary disease (COPD), pulmonary fibrosis, etc.)
* Chronic renal disease (eg: renal failure)
* Obesity (BMI ≥ 30)
* Progressive cancer under treatment
* Chronic haematological pathology
* Chronic liver disease (eg: cirrhosis)
* HIV infection / other immune deficiency (congenital or acquired immunosuppression)
* Has received an organ or bone marrow transplant
* Chronic neurological abnormality / disease
* Immunosuppression
* Subject having his 2nd injection of COVID-19 vaccine scheduled during the 3 weeks of study follow-up
* Taking part in another interventional clinical trial or in the exclusion period to another study
* Those who do not have access to email/internet
* Not capable of giving informed consent
* Hypersensitivity or known allergy to any component of the product
* Patient with a member of his household already included in the study
* Patient living in another region than the recruiting laboratory

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
number of days until resolution of nasal symptoms | From Day 0 to Day 21
  the number of days until resolution of nasal symptoms (nasal obstruction or rhinorrhea) based on the Wisconsin Upper Respiratory Symptom Survey - 21 (WURSS-21) self-questionnaire modified for COVID-19 symptoms.

SECONDARY OUTCOMES:
Symptom resolution | From Day 0 to Day 21
  the number of days until resolution of COVID-19 and URTIs-induced individual symptoms based on the Wisconsin Upper Respiratory Symptom Survey - 21 (WURSS-21) self-questionnaire modified for COVID-19 symptoms.
COVID-19 exacerbation | From Day 0 to Day 21
  percent of subjects with evolution towards more severe COVID-19 stage from Day 0 to Day 21 as defined by the NIH COVID-19 Treatment Guidelines classification (Clinical Spectrum of SARS-CoV-2 Infection)
Symptom relief | From Day 0 to Day 21
  • percent of subjects with complete relief from Day 1 to Day 21 based on a 7-point scale: 0 (no relief) to 6 (complete relief).
Viral load evolution | Day 0, Day 3, Day 5, Day 14 and Day 21
  • percent of subjects with negative RT-PCR for SARS-CoV-2 and URTI viruses by Day 3, Day 5, Day 14 & Day 21
Olfactory disorders | From Day 0 to Day 21
  * percent of subjects with recovery from anosmia & smell disorders from Day 0 to Day 21 based on a 0 to 7 severity scale, where 0 = do not have this symptom, and 7 = Severe.
  * percent of subjects with recovery from taste disorders from Day 0 to Day 21 based on a 0 to 7 severity scale, where 0 = do not have this symptom, and 7 = Severe.
Reported illness days & missed days | From Day 0 to Day 21
  * Number of illness days from Day 0 to Day 21 based on the WURSS-21 self-questionnaire modified for COVID-19 symptoms.
  * Reported missed working days from Day 0 to Day 21
  * Reported missed days of activities from Day 0 to Day 21
Concomitant medications | From Day 0 to Day 21
  Number of days of intake of concomitant medications to relieve symptoms from Day 0 to Day 21 Number of concomitant medications used per day to relieve symptoms from Day 0 to Day 21
Transmission within household contacts | From Day 0 to Day 21
  * percent of clinical manifestations of COVID-19 and URTIs in household contacts
  * percent of SARS-CoV-2 positive cases among household contacts within the incubation period and during the 21 days follow-up period based on questionnaires from the WHO "household transmission investigation protocol for 2019-novel coronavirus (COVID-19)"
Health-care-seeking behaviour | From Day 0 to Day 21
  * percent of subjects consulting a HCP due to their COVID-19 and URTI status from Day 0 to Day 21
  * percent of subjects requiring biological or radiological examinations due to COVID-19 and URTI from Day 0 to Day 21
  * percent of hospitalized subjects due to COVID-19 and URTI from Day 0 to Day 21
Compliance to nasal wash | From Day 0 to Day 21
  The following endpoints are only applicable to subjects randomized to the interventional arm of the study:
  * Number of nasal wash/day from Day 0 to Day 21
  * Number of days of use/week from Day 0 to Day 21 Number of subjects using the advised volume/nasal wash from Day 0 to Day 21
Patient satisfaction | at Day 7, Day 14 and Day 21
  The following endpoints are only applicable to subjects randomized to the interventional arm of the study:
  • Product satisfaction (overall satisfaction, overall perceived efficacy) measured at Day 7, Day 14 and Day 21 based on a 5-point scale with 0=Not at all satisfied, and 4=Very satisfied.
Nasal wash tolerance | From Day 0 to Day 21
  The following endpoints are only applicable to subjects randomized to the interventional arm of the study:
  • Self-reported tolerance with nasal wash from Day 0 to Day 21: nasal burning, nasal irritation, nasal itching, nasal bleeding (epistaxis), nasal dryness based on a 7-point scale with 0= no difficulty, and 6=very unacceptable.
Incidence of Adverse Events/Side Effects | From Day 0 to Day 21
  • Adverse Events reported by all subjects from Day 0 to Day 21
  The following endpoint is only applicable to subjects randomized to the interventional arm of the study:
  • Side effects reported by subjects from Day 0 to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Barbara PERNICONI, Principal Investigator
Locations (1):
- Le Carreau, Cergy, France

REFERENCES:
- [Derived] de Gabory L, Vallet S, Naelten G, Raherison-Semjen C. Seawater nasal wash to reduce symptom duration and viral load in COVID-19 and upper respiratory tract infections: a randomized controlled multicenter trial. Eur Arch Otorhinolaryngol. 2024 Jul;281(7):3625-3637. doi: 10.1007/s00405-024-08518-y. Epub 2024 Feb 20. PMID 38376591